CLINICAL TRIAL: NCT00050310
Title: Natural History of Anthrax: A Study of Primary Infected, Recovered, and Exposed (SPoRE) Individuals and Evaluation of AVA Vaccinated Recipients
Brief Title: Natural History of Anthrax: a Study of Primary Infected, Recovered, and Exposed Individuals (SPoRE); and Evaluation of AVA-Vaccinated Recipients
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020110; 02-I-0110
Record Dates: First submitted 2002-12-03; First posted 2002-12-04 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-08-13

CONDITIONS: Anthrax; Bacillus Infections
Keywords: Anthrax; Natural History; Vaccinated Healthy Volunteer
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute Infection (confirmed or suspected): adults and children with acute anthrax infection
- AVA Recipient/Healthy Volunteer: healthy adults who have received AVA vaccine
- Recovered: adults and children in recovering phase of anthrax infection
- Suspected Exposure: adults and children with suspected exposure to anthrax

SUMMARY:
This study will examine pathophysiology and immune response of anthrax in infected or exposed individuals to learn more about the disease symptoms, prevention and response to treatment. In addition, it will evaluate immune response to the anthrax vaccine AVA (Anthrax Vaccine Adsorbed) in healthy, non-infected individuals.

The following individuals may be eligible for this study:

1. People with confirmed or suspected anthrax (inhalational, cutaneous or gastrointestinal, either acute or recovering);
2. People exposed to anthrax who have no clinical symptoms.
3. Healthy people who have not been exposed to anthrax and have been vaccinated with AVA.

Those enrolled in the study will undergo the following tests and procedures.

Infected and exposed individuals:

* Symptomatic participants will have the following clinical procedures if medically necessary:
* a) blood tests for cell counts, chemistries and evidence of anthrax bacteria;
* b) nasal swab to test for evidence of anthrax
* c) chest X-ray;
* d) computed tomography (CT) scan (special X-rays to examine the lungs or abdomen);
* e) echocardiogram to examine the heart
* f) magnetic resonance imaging (MRI), a special imaging test using a magnetic field and radio waves to examine the infected area of skin and soft tissue for patients with cutaneous anthrax.
* All subjects (with or without symptoms) will have the following research procedures:
* a) blood tests to examine immune response to anthrax;
* b) throat swab to test for evidence of anthrax
* c) nasopharyngeal wash to test for anthrax. Water is sprayed into the nostrils and then allowed to drain for collection in a cup;
* d) induced sputum to test for presence of and immune response to anthrax. A mask with a saline mist is placed over the subject s mouth and nose, causing the subject to cough and produce sputum from the lungs. The sputum is collected in a cup this is for individuals 18 and older who do not undergo bronchoscopy, described below.
* Participants 18 years of age and older may have the following optional research procedures:
* a) leukapheresis or plasmapheresis (see description under non-infected, vaccinated individuals above);
* b) lymph node biopsy. A sample of lymph node tissue is surgically removed under local anesthetic;
* c) bronchoalveolar lavage. This 15- to 30-minute procedure is done in the intensive care unit. The mouth, nasal passages, throat and airways are numbed with lidocaine and a thin flexible tube is passed through the nose into the lung airways. Samples of cells and secretions are obtained by rinsing (lavage) the airways with salt water. The fluid is analyzed for infection, inflammatory cells and inflammatory chemicals.

All infected and exposed individuals will have periodic medical history and physical exam evaluations and be offered treatment or prophylaxis (treatment to prevent infection) with antibiotics, according to the guidelines of the Centers for Disease Control and Prevention (CDC). Patients will be monitored for at least 24 months after antibiotic treatment, or longer if circumstances warrant.

Non-infected, vaccinated individuals

1. medical history and physical examination
2. blood tests-- between 10 and 50 ml (2-10 teaspoons) of blood will be drawn at a time, and not more than 450 ml will be taken in a 6-week period. Based on the blood test results, other optional research procedures may be requested
3. leukapheresis to collect white blood cells and plasmapheresis to collect plasma (the liquid part of the blood). For both of these procedures, blood is collected through a needle placed in an arm vein. The blood flows into a special machine that separates it into its components by spinning. The desired components (white cells or plasma) are removed and the rest of the blood is returned to the body through the same needle or a second needle in the other arm.

DETAILED DESCRIPTION:
The intentional use of Bacillus anthracis in 2001 as a bioterrorism weapon with fatal consequences renewed interest in past epidemiologic and animal research about pathogenesis and posed new dilemmas about diagnosis and treatment. Cases in the October 2001 US outbreak were theoretically exposed via one dispersal method: aerosolization of Ames strain spores. While some developed the cutaneous anthrax form, others sustained the more serious inhalational disease. Inhaled spores are known to travel to alveolar macrophages and then onto the mediastinal lymph nodes where germination to the bacterium form and toxin release are thought to occur. Infective dose, significance of dormant spores after long-term antibiotic therapy, spectrum of disease and even precise cause of death remain unknown. This observational, prospective natural history study was developed during the 2001 outbreak and is set up to follow participants from the time of exposure through post-recovery (greater than ten years). Healthy vaccinated participants have been included to evaluate serum titers and cell markers in relation to dose and frequency of Anthrax Vaccine Adsorbed (AVA) vaccine.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects at least 3 years old, including pregnant women, are eligible for inclusion if they meet one of the five criteria listed below, are hemodynamically and clinically stable, and agree to stored samples. Women of child-bearing age or potential will not be excluded from participation but pregnancy status will be determined by serum or urine pregnancy test at time of enrollment in order to optimize subsequent evaluation and care.

Although the study is open to participants at least 3 years old, pediatric anthrax cases are historically rare and essentially of the cutaneous type. Therefore, few, if any pediatric subjects are expected.

Decisionally impaired subjects will be included in this study only if a Legally Authorized Representative (LAR) understands and is willing to sign a written informed consent document.

1. Inhalation Anthrax (acute or recovering infection)

   CONFIRMED:

   --nonspecific febrile illness followed by sepsis and/or respiratory failure

   AND

   --B anthracis isolation (via culture) from any site OR 2 supportive lab tests

   OR SUSPECTED:

   --nonspecific febrile illness followed by sepsis and/or respiratory failure with no alternative diagnosis

   AND

   --one supportive lab test OR direct epidemiological link to a confirmed environmental exposure
2. Cutaneous Anthrax (acute or recovering infection)

   CONFIRMED:

   --characteristic lesion (papule->vesicular->depressed black eschar plus or minus edema, erythema, necrosis, or ulceration)

   AND

   --B anthracis isolation (culture) from any site OR 2 supportive lab tests

   SUSPECTED:

   --Characteristic lesion with no alternative diagnosis

   AND

   --one supportive lab test OR direct epidemiological link to a confirmed environmental exposure
3. Gastrointestinal Anthrax (acute or recovering infection)

   CONFIRMED:

   --Severe abdominal pain often associated with bloody vomiting/diarrhea followed by fever/septicemia

   AND

   --B anthracis isolation (culture) from any site OR 2 supportive lab tests

   SUSPECTED:

   --Severe abdominal pain often associated with bloody vomiting/diarrhea followed by fever/septicemia with no alternative diagnosis

   AND

   --1 supportive lab test OR direct epidemiological link to a confirmed environmental exposure

   These definitions were subsequently updated by the CDC in 2010 to accept clinically compatible symptoms plus one of the following: a positive culture, a positive immunohistochemical stain for antigen, a 4-fold increase in anti-PA IgG or a positive documented exposure with detection of DNA via PCR (26).
4. Exposed individuals who are clinically asymptomatic.
5. Past or imminent vaccination in healthy (non-anthrax exposed).
6. Hemodynamically and clinically stable at time of evaluation at NIH.

   * Hemodynamically: stable vital signs
   * Clinically: no obvious signs of disease progression (e.g. worsening pleural effusions or increasing cutaneous edema)
   * acute/newly recovered patients must be receiving standard antimicrobial therapy
7. Participant agrees to stored samples.

EXCLUSION CRITERIA:

Inability of subject or Legally Authorized Representative (LAR) to understand or subject not willing to sign a written informed consent document.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have recovered from anthrax infection. Cohorts are based on route of infection.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2002-10-31 (Actual)

PRIMARY OUTCOMES:
evaluate the natural history of anthrax and immune response to anthrax antigens over time | 2 years
  This study is intended to evaluate the natural history of anthrax and the immune response to anthrax over time in four subpopulations of men, women and children with: --acute infection (confirmed or suspected) --recovering phase of infection --exposure to infection --no known or no exposure to infection but a history of anthrax vaccination (AVA) (since no children have received AVA, they will be excluded from this subgroup)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Wright, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dalton R. Genetic sleuths rush to identify anthrax strains in mail attacks. Nature. 2001 Oct 18;413(6857):657-8. doi: 10.1038/35099687. No abstract available. PMID 11606978
- [Background] Shafazand S, Doyle R, Ruoss S, Weinacker A, Raffin TA. Inhalational anthrax: epidemiology, diagnosis, and management. Chest. 1999 Nov;116(5):1369-76. doi: 10.1378/chest.116.5.1369. PMID 10559102
- [Background] Centers for Disease Control and Prevention (CDC). Update: Investigation of bioterrorism-related anthrax and adverse events from antimicrobial prophylaxis. MMWR Morb Mortal Wkly Rep. 2001 Nov 9;50(44):973-6. PMID 11724150
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-I-0110.html